CLINICAL TRIAL: NCT01846299
Title: A 12-month, Randomized, Double-masked, Sham-controlled, Multicenter Study to Evaluate the Efficacy and Safety of 0.5mg Ranibizumab Intravtitreal Injections in Patients With Visual Impairment Due to Vascular Endothelial Growth Factor (VEGF)Driven Macular Edema
Brief Title: To Assess the Efficacy and Safety of Intravitreal Ranibizumab in People With Vision Loss Due to Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRFB002G2302; 2012-005418-20 (EudraCT Number)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Macular Edema (ME)
Keywords: Vision Impairment
MeSH Terms: conditions — Macular Edema; Vision Disorders | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Experimental): A 0.5 mg ranibizumab intravitreal injection was given to the study eye at baseline, and then as needed based on evidence of disease activity.
  Interventions: Drug: Ranibizumab
- Sham control (Sham Comparator): Sham injection was given to the study eye at baseline, and then treatment was given based on evidence of disease activity. At month 1, if treatment was needed, sham was administered. At month 2, participants switched to open-label ranibizumab on an as needed basis.
  Interventions: Other: Sham control

INTERVENTIONS:
Other: Sham control — The sham vial did not contain active drug (empty sterile vial). The sham injection was an imitation of an intravitreal injection using an injection syringe without a needle touching the eye.
  Arms: Sham control
Drug: Ranibizumab — Ranibizumab 0.5mg/0.5mL was administered intravitreally to the participant.
  Arms: Ranibizumab

SUMMARY:
To evaluate the efficacy and safety of 0.5 mg Ranibizumab intravitreal injections in adult patients with visual impairment due to macular edema (ME).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active ME secondary to any causes (for adult patients: except diabetic macular edema (DME), age-related macular degeneration (AMD) and retinal vein occlusion (RVO));
* BCVA must be between ≥ 24 and ≤ 83 letters;
* Visual loss should be mainly due to the presence of any eligible types of ME.

Exclusion Criteria:

* Women of child-bearing potential,
* Active malignancies;
* History of stroke less than 6 months prior to screening;
* Uncontrolled systemic inflammation or infection, related directly to the underlying causal disease of ME;
* Active diabetic retinopathy, active ocular/periocular infectious disease or active severe intra-ocular inflammation;
* Any type of advanced, severe or unstable ocular disease or its reatment;
* ME with a high likelihood of spontaneous resolution.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- Australia (5):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, South Launceston, Tasmania
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Halifax, Nova Scotia, Canada
- Czechia (2):
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- France (4):
  - Novartis Investigative Site, Bordeaux, France
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Jean
- Germany (4):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Regensburg, Germany
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg I. Br
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Israel (5):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (6):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Riga, Latvia
- Netherlands (2):
  - Novartis Investigative Site, Tilburg, Netherlands
  - Novartis Investigative Site, Amsterdam
- Russia (2):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica, Slovakia
  - Novartis Investigative Site, Trenčín, Slovakia
- South Korea (3):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
- Switzerland (3):
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Binningen
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Kocaeli
- United Kingdom (7):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Sunderland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 181 participants were enrolled. Of these, 178 adults were randomized in a 2:1 ratio and considered for analysis. The 3 adolescent participants, non-randomized, received open-label treatment and were not included in the analyses. Therefore, the number enrolled = 181 differs from the number randomized = 178 in the participant flow.
Groups:
- Sham: Sham injection was given to the study eye at baseline, and then treatment was given based on evidence of disease activity. At Month 1, if treatment was needed, sham was administered. At Month 2, participants could switch to open-label ranibizumab on an as needed basis.
Period: Overall Study
Arm/Group | Ranibizumab | Sham
Started | 118 | 60
Full Analysis Set | 117 (One participant did not receive study treatment prior to discontinuation.) | 60
Safety Set | 119 (Two participants randomized to sham received ranibizumab at Month 1.) | 58
Completed | 106 | 50
Not Completed | 12 | 10
Not completed — Physician Decision | 4 | 2
Not completed — Protocol deviation | 1 | 0
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Sham | Total
Number analyzed (Participants) | 118 | 60 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (13.97) | 61.8 (15.55) | 62.9 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 23 | 68
  Male | 73 | 37 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) in Study Eye
Description: BCVA was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity (VA) testing charts at an initial testing distance of 4 meters. A positive change from baseline indicated improvement.
Time Frame: Baseline, Month 2
Population: Full analysis set: The full analysis set included all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: letters
Groups:
- Sham With Ranibizumab: Sham injection was given to the study eye at baseline, and then treatment was given based on evidence of disease activity. At Month 1, if treatment was needed, sham was administered. At Month 2, participants could switch to open-label ranibizumab on an as needed basis.
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
letters | 5.7 (0.81) | 2.9 (0.89)
Statistical Analysis 1: Comparison: Ranibizumab vs Sham With Ranibizumab; Test type: Superiority or Other; p = 0.0111, Mixed Models Analysis; Mean Difference (Net) = 2.78, 95% CI 2-sided [0.40 to 5.16], Standard Error of Mean 1.203

2. Secondary Outcome: Change From Baseline in BCVA in Study Eye up to Month 2
Description: as for outcome 1
Time Frame: Baseline, Month 1, Month 2
Population: The full analysis set (FAS) was considered for the analysis. The FAS. The FAS included all randomized participants who received at least one dose of study treatment. Only participants of the FAS, who had data at baseline and the specific post-baseline time point, were included in the analysis for that time point.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
letters
  Month 1 (n=116,59) | 4.7 (0.70) | 1.4 (0.98)
  Month 2 (n=114,59) | 5.8 (0.76) | 2.8 (1.05)

3. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CSFT) in Study Eye
Description: CSFT wasassessed by optical coherence tomography (OCT). A negative change from baseline indicates improvement.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: The full analysis set (FAS) was considered for the analysis. The FAS included all randomized participants who received at least one dose of study treatment. Only participants of the FAS, who had data at baseline and the specific post-baseline time point, were included in the analysis for that time point.
Measure: Mean (Standard Deviation); unit: micrometers (um)
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
micrometers (um)
  Month 1 (n=112,59) | -83.6 (127.45) | -14.3 (97.36)
  Month 2 (n=112,59) | -82.5 (140.06) | -30.6 (102.77)
  Month 3 (n=113,59) | -86.5 (136.43) | -92.2 (129.85)
  Month 4 (n=109,57) | -94.5 (141.55) | -95.5 (140.68)
  Month 5 (n=105,57) | -98.6 (136.28) | -107.6 (142.22)
  Month 6 (n=109,54) | -110.6 (133.10) | -84.1 (137.86)
  Month 7 (n=105,52) | -113.3 (130.84) | -112.9 (148.13)
  Month 8 (n=105,51) | -113.1 (127.11) | -107.7 (157.40)
  Month 9 (n=105,52) | -111.6 (127.99) | -116.3 (146.43)
  Month 10 (n=103,50) | -114.1 (131.12) | -116.6 (147.26)
  Month 11 (n=101,49) | -112.1 (124.00) | -123.5 (140.65)
  Month 12 (n=103,50) | -121.0 (124.67) | -116.8 (137.99)

4. Secondary Outcome: Change From Baseline in Central Subfield Volume (CSFV) in Study Eye
Description: CSFV was assessed OCT. A negative change from baseline indicates improvement.
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microliters (ul)
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
microliters (ul)
  Month 1 (n=112,59) | -0.296 (0.4570) | -0.032 (0.3969)
  Month 2 (n=112,59) | -0.276 (0.5362) | -0.104 (0.3958)
  Month 3 (n=113,59) | -0.322 (0.5812) | -0.348 (0.5075)
  Month 4 (n=109,57) | -0.333 (0.5568) | -0.378 (0.5436)
  Month 5 (n=105,57) | -0.383 (0.5592) | -0.401 (0.5893)
  Month 6 (n=109,54) | -0.388 (0.5167) | -0.344 (0.5530)
  Month 7 (n=105,52) | -0.438 (0.5267) | -0.438 (0.6098)
  Month 8 (n=105,51) | -0.405 (0.5074) | -0.421 (0.6484)
  Month 9 (n=105,52) | -0.446 (0.6066) | -0.444 (0.6210)
  Month 10 (n=103,50) | -0.439 (0.6241) | -0.433 (0.6407)
  Month 11 (n=101,49) | -0.406 (0.4871) | -0.459 (0.6157)
  Month 12 (n=103,50) | -0.447 (0.4837) | -0.455 (0.5910)

5. Secondary Outcome: Number of Participants With Presence or Absence of Intra-retinal Fluid in Study Eye Compared to Baseline
Description: The presence of intra-retinal fluid was assessed by OCT.
Time Frame: Month 2, Month 6, Month 12
Population: The FAS was considered for the analysis. The FAS included all randomized participants who received at least one dose of study treatment. Only participants (n), with values 'Absent' or 'Definite' for both the baseline and corresponding post-baseline time point, were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
Participants
  Month 2, Absent (n=112,59) | 98 | 46
  Month 2, Definite (n=112,59) | 14 | 13
  Month 6, Absent (n=109,55) | 97 | 43
  Month 6, Definite (n=109,55) | 12 | 12
  Month 12, Absent (n=103,50) | 78 | 39
  Month 12, Definite (n=103,50) | 25 | 11

6. Secondary Outcome: Number of Participants With Presence or Absence of Subretinal Fluid in Study Eye Compared to Baseline
Description: The presence of subretinal fluid was assessed by OCT.
Time Frame: Month 2, Month 6, Month 12
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
Participants
  Month 2, Absent (n=113,59) | 77 | 33
  Month 2, Definite (n=110,55) | 36 | 26
  Month 6, Absent (n=109,55) | 75 | 35
  Month 6, Definite (n=109,55) | 35 | 20
  Month 12, Absent (n=104,50) | 77 | 37
  Month 12, Definite (n=103,50) | 27 | 13

7. Secondary Outcome: Number of Participants With Presence of Active Macular Edema (ME) Leakage
Description: The presence of active ME leakage was assessed by fluorescein angiography (FA).
Time Frame: Month 2
Population: The FAS was used this analysis. The FAS included randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
Participants | 96 | 53

8. Secondary Outcome: Number of Participants Requiring Rescue Treatment at Month 1
Description: Rescue treatment with laser photocoagulation or periocular treatment could be administered at Month 1 only if the participant had a visual acuity loss of > 5 letters due to disease activity from baseline to Month 1.
Time Frame: Month 1
Population: The FAS was used for this analysis. The FAS included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
Participants | 0 | 0

9. Secondary Outcome: Average Change From Baseline in BCVA
Description: as for outcome 1
Time Frame: Baseline (BL), month 1 through month 6, month 1 through month 12
Population: The FAS was used for this analysis. The FAS included randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
letters
  Average change from BL, month 1 through month 6 | 6.39 (8.405) | 4.50 (8.095)
  Average change from BL, month 1 through month 12 | 7.40 (9.052) | 5.82 (8.927)

10. Secondary Outcome: Number of Participants With ≥ 1, ≥ 5, ≥ 10 and ≥ 15 Letters Gain or Reaching 84 Letters
Description: VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using ETDRS-like visual acuity testing charts at a testing distance of 4 meters.
Time Frame: Month 2, Month 6 , Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
Participants
  Month 2, Gain of >= 15 letters (n=114,59) | 26 | 7
  Month 2, Gain of >= 10 letters (n=114,59) | 35 | 11
  Month 2, Gain of >= 5 letters (n=114,59) | 55 | 19
  Month 2, Gain of >= 1 letter (n=114,59) | 80 | 38
  Month 6, Gain of >= 15 letters (n=111,55) | 30 | 15
  Month 6, Gain of >= 10 letters (n=111,55) | 41 | 21
  Month 6, Gain of >= 5 letters (n=111,55) | 67 | 34
  Month 6, Gain of >= 1 letters (n=111,55) | 87 | 40
  Month 12, Gain of >= 15 letters (n=106,50) | 44 | 22
  Month 12, Gain of >= 10 letters (n=106,50) | 55 | 27
  Month 12, Gain of >= 5 letters (n=106,50) | 72 | 37
  Month 12, Gain of >= 1 letters (n=106,50) | 86 | 42

11. Secondary Outcome: Number of Participants With > 1, > 5, > 10 and > 15 Letters Loss
Description: as for outcome 10
Time Frame: Month 2, Month 6, Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab
Number analyzed (Participants) | 117 | 60
Participants
  Month 2, Loss of >1 letter (n=114,59) | 17 | 9
  Month 2, Loss of >5 letters (n=114,59) | 8 | 4
  Month 2, Loss of >10 letters (n=114,59) | 2 | 3
  Month 2, Loss of >15 letters (n=114,59) | 0 | 0
  Month 6, Loss of >1 letter (n=111,55) | 14 | 12
  Month 6, Loss of >5 letters (n=111,55) | 5 | 7
  Month 6, Loss of >10 letters (n=111,55) | 3 | 4
  Month 6, Loss of >15 letters (n=111,55) | 1 | 1
  Month 12, Loss of >= 1 letter (n=106,50) | 10 | 5
  Month 12, Loss of >= 5 letters (n=106,50) | 6 | 3
  Month 12, Loss of >= 10 letters (n=106,50) | 2 | 3
  Month 12, Loss of >= 15 letters (n=106,50) | 1 | 2

12. Secondary Outcome: Number of Participants With Ranibizumab Treatments
Description: The number of participants administered study treatments, according to treatment frequency, was assessed.
Time Frame: Month 12
Population: The safety set was used for this analysis. The safety set included randomized participants who received at least one dose of study treatment. Two participants from the sham group were included in the ranibizumab group based on the actual treatment received.
Measure: Number; unit: Participants
Groups:
- Sham Without Ranibizumab: Participants did not receive ranibizumab at any time during the study.
Arm/Group | Ranibizumab | Sham With Ranibizumab | Sham Without Ranibizumab
Number analyzed (Participants) | 119 | 56 | 2
Participants
  Frequency of injections = 0 | 0 | 0 | 2
  Frequency of injections = 1 | 13 | 6 | 0
  Frequency of injections = 2 | 5 | 3 | 0
  Frequency of injections = 3 | 14 | 7 | 0
  Frequency of injections = 4 | 3 | 5 | 0
  Frequency of injections = 5 | 17 | 7 | 0
  Frequency of injections = 6 | 7 | 11 | 0
  Frequency of injections = 7 | 6 | 0 | 0
  Frequency of injections = 8 | 13 | 0 | 0
  Frequency of injections = 9 | 3 | 6 | 0
  Frequency of injections = 10 | 12 | 11 | 0
  Frequency of injections = 11 | 6 | 0 | 0
  Frequency of injections = 12 | 20 | 0 | 0

13. Secondary Outcome: Number of Participants With Re-treatments
Description: The number of participants, administered re-treatments according to treatment frequency, was assessed. Re-treatment was defined as an administration of study medication following at least one non-missed visit where treatment was not administered in the study eye. Up to Month 12, the maximum number of retreatments was 5.
Time Frame: Month 6, month 12
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham With Ranibizumab | Sham Without Ranibizumab
Number analyzed (Participants) | 119 | 56 | 2
Participants
  Month 6, Frequency of re-treatment = 1 | 34 | 15 | 0
  Month 6, Frequency of re-treatment = 2 | 15 | 3 | 0
  Month 12, Frequency of re-treatment = 1 | 21 | 12 | 0
  Month 12, Frequency of re-treatment = 2 | 24 | 7 | 0
  Month 12, Frequency of re-treatment = 3 | 13 | 5 | 0
  Month 12, Frequency of re-treatment = 4 | 5 | 5 | 0
  Month 12, Frequency of re-treatment = 5 | 3 | 0 | 0

14. Secondary Outcome: Number of Primary Reasons for Decision to Treat by Investigator
Description: The total number of primary reasons for decisions to treat was assessed. A single participant could have had multiple primary reasons for treatment.
Time Frame: 12 months
Population: as for outcome 12
Measure: Number; unit: Number of primary reasons
Units Other Than Participants: Reasons
Arm/Group | Ranibizumab | Sham With Ranibizumab | Sham Without Ranibizumab
Number analyzed (Participants) | 119 | 56 | 2
Number analyzed (Reasons) | 689 | 372 | 1
Number of primary reasons
  Vision impairment | 38 | 22 | 0
  OCT abnormality | 637 | 345 | 1
  FA abnormality | 11 | 5 | 0
  Color fundus photography abnormality | 0 | 0 | 0
  Clinical abnormality | 3 | 0 | 0
  Without documentation (missing reason) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Ranibizumab 0.5mg: Ranibizumab 0.5mg
- Sham With Ranibizumab 0.5mg: Sham with Ranibizumab 0.5mg
- Sham Without Ranibizumab 0.5mg: Sham without Ranibizumab 0.5mg
Arm/Group | Ranibizumab 0.5mg | Sham With Ranibizumab 0.5mg | Sham Without Ranibizumab 0.5mg
Serious Adverse Events (participants affected / at risk) | 15/119 | 6/56 | 1/2
Other Adverse Events (participants affected / at risk) | 58/119 | 21/56 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg (N=119) | Sham With Ranibizumab 0.5mg (N=56) | Sham Without Ranibizumab 0.5mg (N=2)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Conjunctivitis allergic (Fellow treated eye) (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Study eye) (Eye disorders) | 1 | 0 | 0
Corneal oedema (Fellow treated eye) (Eye disorders) | 0 | 1 | 0
Open angle glaucoma (Fellow untreated eye) (Eye disorders) | 1 | 0 | 0
Open angle glaucoma (Study eye) (Eye disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Endophthalmitis (Study eye) (Infections and infestations) | 1 | 0 | 0
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 0 | 0 | 1
Brain stem stroke (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg (N=119) | Sham With Ranibizumab 0.5mg (N=56) | Sham Without Ranibizumab 0.5mg (N=2)
Conjunctival haemorrhage (Study eye) (Eye disorders) | 11 | 7 | 0
Cystoid macular oedema (Study eye) (Eye disorders) | 6 | 0 | 0
Dry eye (Study eye) (Eye disorders) | 6 | 1 | 0
Eye pain (Study eye) (Eye disorders) | 10 | 2 | 0
Macular oedema (Fellow untreated eye) (Eye disorders) | 1 | 3 | 0
Macular oedema (Study eye) (Eye disorders) | 7 | 2 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 11 | 3 | 0
Influenza (Infections and infestations) | 6 | 3 | 0
Nasopharyngitis (Infections and infestations) | 12 | 2 | 0
Intraocular pressure increased (Study eye) (Investigations) | 6 | 3 | 0
Hypertension (Vascular disorders) | 6 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.